CLINICAL TRIAL: NCT01360658
Title: Phase 2 Multicentric Study Evaluating the Efficacy of Polyvalent Intravenous Immunoglobulins in Idiopathic Severe and Refractory Solar Urticaria
Brief Title: Intravenous Immunoglobulins in Severe and Refractory Solar Urticaria
Acronym: IGUS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Ministry of Health, France (Other Government); Saint-Louis Hospital, Paris, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N/2010/57
Record Dates: First submitted 2011-05-23; First posted 2011-05-25 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Solar Urticaria
Keywords: Intravenous immunoglobulins; Solar urticaria; Minimal urticaria dose; Quality of life; Safety
MeSH Terms: conditions — Urticaria, Solar | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intravenous immunoglobulins (Experimental): Intravenous immunoglobulins
  Interventions: Drug: Intravenous immunoglobulins

INTERVENTIONS:
Drug: Intravenous immunoglobulins — Single administration of 2 g/kg intravenous immunoglobulins over 2 days
  Other Names: CLAIRYG

SUMMARY:
Solar urticaria is a rare but debilitating disease that can severely impact the quality of life, restricting outdoor activities.Treatment, based on sun protection and anti-histaminic drugs, is efficacious in 2 patients out of 3. In refractory patients, photodesensitization or immunosuppressive treatments such as cyclosporin A can be proposed. As in idiopathic urticaria, intravenous immunoglobulins (IVIG)have been shown, in a retrospective study of 7 patients, to dramatically improve 71% of patients. In an open-label prospective multicenter study, we aim to demonstrate the efficacy of a single IVIG administration (2g/kg) in 10 patients affected with severe and refractory solar urticaria.

ELIGIBILITY:
Inclusion Criteria:

* social insurance
* signed informed consent
* solar urticaria (SU) confirmed with photoexplorations
* SU involving the face or generalized to the whole body or accompanied with bronchospasm or triggered by artificial light or per annual SU
* SU with altered quality of life
* SU resistant to photoprotection
* SU resistant to the association of two different antihistaminics during 3 months

Exclusion Criteria:

* Pregnancy
* Heat triggered urticaria
* Contra-indications to IVIG

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Percentage of patients obtaining 3 months after treatment a 10 fold increase of pretherapeutic minimal urticarial dose | 3 months

SECONDARY OUTCOMES:
Percentage of patients obtaining 1 month after treatment a 10 fold increase of pretherapeutic minimal urticarial dose | 1 month
Percentage of patients obtaining 1 month after treatment an improvement of quality of life | 1 month
Percentage of patients obtaining after 1 month of treatment a complete clinical response | 1 month
Percentage of patients obtaining 1 month after treatment a 50% and a 75% improvement of disease severity | 1 month
Percentage of patients obtaining 6 months after treatment a 10 fold increase of pretherapeutic minimal urticarial dose | 6 months
Percentage of patients obtaining 12 months after treatment a 10 fold increase of pretherapeutic minimal urticarial dose | 12 months
Percentage of patients obtaining 3 months after treatment an improvement of quality of life | 3 months
Percentage of patients obtaining 6 months after treatment an improvement of quality of life | 6 months
Percentage of patients obtaining 12 months after treatment an improvement of quality of life | 12 months
Percentage of patients obtaining after 3 months of treatment a complete clinical response | 3 months
Percentage of patients obtaining after 6 months of treatment a complete clinical response | 6 months
Percentage of patients obtaining after 12 months of treatment a complete clinical response | 12 months
Percentage of patients obtaining 3 months after treatment a 50% and a 75% improvement of disease severity | 3 months
Percentage of patients obtaining 6 months after treatment a 50% and a 75% improvement of disease severity | 6 months
Percentage of patients obtaining 12 months after treatment a 50% and a 75% improvement of disease severity | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: François Aubin, Pr, Principal Investigator — University Hospital of Besançon; Manuelle Viguier, Dr, Principal Investigator — Saint-Louis Hospital, Paris, France
Locations (12):
- France (12):
  - Regional University Hospital, Besançon
  - University Hospital, Caen
  - University Hospital, Grenoble
  - Regional University Hospital, Lille
  - University hospital, Limoges
  - Regional University Hospital, Montpellier
  - University Hospital, Nancy
  - University Hospital, Nîmes
  - Saint louis Hospital, Paris
  - University Hospital, Reims
  - University Hospital, Rennes
  - University Hospital, Toulouse